CLINICAL TRIAL: NCT03535844
Title: Cardio-vascular Protective Effects of Wolfberry in Middle-aged and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other); Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S2
Record Dates: First submitted 2018-04-22; First posted 2018-05-24 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases; Aging
Keywords: Wolfberry (Goji berry); Healthy diet; Cardiovascular diseases; Endothelial function; Lipidomics; Middle-aged and older adults; Oxidative stress; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wolfberry with healthy diet (Experimental): Each subject will be provided one-to-one dietary counselling by a research dietitian and an instruction sheet to achieve the healthy eating pattern diet. Subjects will also be provided specific instructions to cook and consume 15 g/day wolfberry as part of a mixed-meal.
  Interventions: Other: Wolfberry; Other: Healthy diet
- Healthy diet (Active Comparator): Each subject will be provided one-to-one dietary counselling by a research dietitian and an instruction sheet to achieve the healthy eating pattern diet.
  Interventions: Other: Healthy diet

INTERVENTIONS:
Other: Wolfberry — Consumption of cooked dehydrated wolfberry as part of a mixed meal.
  Arms: Wolfberry with healthy diet
Other: Healthy diet — Compliance to a healthy diet in accordance to recommendations by the Singapore Health Promotion Board.

SUMMARY:
This purpose of this study is to assess the impact of consuming wolfberry on cardiovascular risk in Singapore's middle-aged and older adults. The investigators hypothesize that consuming wolfberry with a healthy eating pattern diet will contribute to improvements in cardiovascular health when compared to a similar diet without wolfberry.

DETAILED DESCRIPTION:
This is a 16-week parallel, single-blind (investigator), prospective randomized controlled trial. The study was designed based on previous research which showed that consuming 15 g/day of wolfberry for 4 weeks and 14 g/day of wolfberry with meal for 6 weeks increased plasma zeaxanthin concentrations and antioxidant status. Also, other studies reported observable changes in the endothelial progenitor cells and flow mediated dilation after just two weeks of fruit and vegetables or healthy diet interventions. Thus collectively, 16-weeks may be a sufficient period to detect the changes in endothelial function, whole body carotenoids, and anti-oxidant status, which are the outcomes of interest in this research project.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give an informed consent
2. Age 50 to 75 years
3. Willing to follow the study procedures

Exclusion Criteria:

1. Significant change in weight (± 5% body weight) during the past 3 months
2. Allergy to wolfberry
3. Acute illness at the study baseline
4. Exercising vigorously over the past 3 months
5. Consistently following healthy eating pattern diet in the past 3 months
6. Smoking
7. Have an average weekly alcohol intake that above 21 units per week (males) and 14 units per week (females): 1 unit = 360 mL of beer; 150 mL of wine; 45 mL of distilled spirits)
8. Pregnant, lactating, or planning pregnancy in the next 6 months
9. Taking dietary supplements which may impact the outcome of interests (e.g. vitamin supplements, antioxidant supplement etc.)
10. Prescribed and taking antihypertensive/cholesterol-lowering/ type-2 diabetic medication which started less than 5 years prior to the intervention participation
11. Insufficient venous access to allow the blood collection

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, PhD, RD, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University of Singapaore, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure website with access limited to the principal investigator and her research staff. All data will be de-identified prior to statistical analyses

REFERENCES:
- [Background] de Souza Zanchet MZ, Nardi GM, de Oliveira Souza Bratti L, Filippin-Monteiro FB, Locatelli C. Lycium barbarum Reduces Abdominal Fat and Improves Lipid Profile and Antioxidant Status in Patients with Metabolic Syndrome. Oxid Med Cell Longev. 2017;2017:9763210. doi: 10.1155/2017/9763210. Epub 2017 Jun 8. PMID 28685012
- [Background] Cheng CY, Chung WY, Szeto YT, Benzie IF. Fasting plasma zeaxanthin response to Fructus barbarum L. (wolfberry; Kei Tze) in a food-based human supplementation trial. Br J Nutr. 2005 Jan;93(1):123-30. doi: 10.1079/bjn20041284. PMID 15705234
- [Derived] Toh DWK, Xia X, Sutanto CN, Low JHM, Poh KK, Wang JW, Foo RS, Kim JE. Enhancing the cardiovascular protective effects of a healthy dietary pattern with wolfberry (Lycium barbarum): A randomized controlled trial. Am J Clin Nutr. 2021 Jul 1;114(1):80-89. doi: 10.1093/ajcn/nqab062. PMID 33964853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Started | 22 | 19
Completed | 22 | 18
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Apparently healthy middle-aged and older adults in Singapore
Groups:
- Total: Total of all reporting groups
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (4) | 56 (4) | 56 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 17 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 22 | 18 | 40
Use of prescription medication and/or supplements [Count of Participants; unit: Participants] | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Lipidomic Profiles
Description: The main classes of lipids in the cell membrane
Time Frame: Pre- and post-intervention (Week 16)
Reporting Status: Not Posted, anticipated posting 2020-09

2. Primary Outcome: Change in Carotid Intima Media Thickness
Description: Carotid intima media thickness measured using high-frequency ultrasonographic imaging
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
mm
  Week 0 | 0.67 (0.11) | 0.60 (0.10)
  Week16 | 0.67 (0.12) | 0.70 (0.09)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.49, t-test, 2 sided; independent t-test of change values
Statistical Analysis 2: Comparison: Healthy Diet; Test type: Superiority; p = 0.5672, t-test, 1 sided; Paired t-test (Week 0 and Week 16)
Statistical Analysis 3: Comparison: Wolfberry With Healthy Diet; Test type: Superiority; p = 0.788, t-test, 2 sided; Paired t-test of change values

3. Primary Outcome: Change in Endothelial Progenitor Cells
Description: Quantity and quality of circulating endothelial progenitor cells
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
cells
  Week 0 | 9.89 (3.43) | 10.36 (2.67)
  Week 16 | 9.64 (2.29) | 9.46 (2.87)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.67, t-test, 2 sided; independent t-test of change values
Statistical Analysis 2: Comparison: Healthy Diet; Test type: Superiority; p = 0.8203, t-test, 2 sided; Paired t-test of change values
Statistical Analysis 3: Comparison: Wolfberry With Healthy Diet; Test type: Superiority; p = 0.3882, t-test, 2 sided; Paired t-test of change values

4. Primary Outcome: Change in Flow Mediated Dilation
Description: Brachial artery flow mediated dilation measured using high-frequency ultrasonographic imaging
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: % dilation
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
% dilation
  Week 0 | 4.50 (3.24) | 3.95 (3.12)
  Week 16 | 3.79 (2.68) | 5.34 (2.49)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.08, t-test, 2 sided; independent t-test of change values

5. Primary Outcome: Change in Plasma Nitric Oxide
Description: Concentrations of plasma total nitrate/nitrite using commercially available ELISA assay kits.
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
nmol/mL
  Nitric oxide Week 0 | 15.91 (8.39) | 14.53 (6.8)
  Nitric oxide Week 16 | 19.38 (10.12) | 19.55 (8.27)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.7162, t-test, 2 sided; independent t-test of change values
Statistical Analysis 2: Comparison: Healthy Diet; Test type: Superiority; p = 0.07, t-test, 2 sided; Paired t-test of Week 0 and Week 16 nitric oxide values
Statistical Analysis 3: Comparison: Wolfberry With Healthy Diet; Test type: Superiority; p < 0.05, t-test, 2 sided; Paired t-test of Week 0 and Week 16 nitric oxide values

6. Primary Outcome: Change in Blood Carotenoid Status
Description: Fasting state plasma carotenoids using high performance liquid chromatography.
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
nmol/L
  Week 0 | 2020.9 (192.3) | 2746.3 (224)
  Week 16 | 1916.2 (218.7) | 1682.9 (209.7)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p < 0.05, t-test, 2 sided; Independent t-test of change values

7. Secondary Outcome: Change in Blood Lipid-lipoprotein Concentrations
Description: Total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and total triglyceride
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
mmol/L
  TG Week 0 | 1.18 (0.54) | 1.32 (0.62)
  TG Week 16 | 1.15 (0.52) | 1.36 (0.73)
  TC Week 0 | 5.16 (0.87) | 5.36 (1.17)
  TC Week 16 | 5.30 (0.88) | 5.31 (1.16)
  LDL Week 0 | 3.06 (0.63) | 3.23 (1.10)
  LDL Week 16 | 3.14 (0.6) | 3.16 (1.11)
  HDL Week 0 | 1.56 (0.49) | 1.54 (0.42)
  HDL Week 16 | 1.65 (0.47) | 1.53 (0.39)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.4855, t-test, 2 sided; Independent t-test of change triglyceride values
Statistical Analysis 2: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.1393, t-test, 2 sided; Independent t-test of change total cholesterol values
Statistical Analysis 3: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.2221, t-test, 2 sided; Independent t-test of change LDL cholesterol values
Statistical Analysis 4: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.078, t-test, 2 sided; Independent t-test of change HDL cholesterol values
Statistical Analysis 5: Comparison: Wolfberry With Healthy Diet; Test type: Superiority; p < 0.05, t-test, 2 sided; Paired t-test of Week 0 and Week 16 HDL cholesterol values
Statistical Analysis 6: Comparison: Healthy Diet; Test type: Superiority; p = 0.7261, t-test, 2 sided; Paired t-test of Week 0 and Week 16 HDL cholesterol values

8. Secondary Outcome: Change in Blood Pressure
Description: Both systolic and diastolic blood pressure
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
mmHg
  Systolic Week 0 | 114 (18) | 106 (13)
  Systolic Week 16 | 111 (15) | 107 (13)
  Diastolic Week 0 | 72 (12) | 69 (9)
  Diastolic Week 16 | 73 (10) | 69 (7)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.1951, t-test, 2 sided; Independent t-test of systolic blood pressure change values
Statistical Analysis 2: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.916, t-test, 2 sided; Independent t-test of diastolic blood pressure change values

9. Secondary Outcome: Change in Oxidative Stress-related Biomarkers
Description: Concentrations of plasma biomarkers of oxidative stress.
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
uM
  MDA Week 0 | 0.294 (0.021) | 0.327 (0.037)
  MDA Week 16 | 0.282 (0.021) | 0.316 (0.025)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.9882, t-test, 2 sided; independent t-test of malondialdehyde change values

10. Secondary Outcome: Change in Body Composition
Description: Dual-energy X-ray absorptiometry
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: % Body Fat
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
% Body Fat
  % Body Fat Week 0 | 36.5 (6.9) | 35.1 (6.1)
  % Body Fat Week 16 | 36.2 (7.4) | 34.4 (7.4)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.4408, t-test, 2 sided; Independent t-test of body fat % change values

11. Secondary Outcome: Change in Skin Carotenoid Status
Description: Measured using resonance Raman spectroscopy to obtain a skin carotenoid status, a score which ranges from 10000 to 89000. Higher score represents higher concentration of carotenoids in skin, hence, an improved outcome
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
score on a scale
  Week 0 | 33636 (2724) | 33713 (1954)
  Week 16 | 37879 (2841) | 35426 (2065)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.1487, t-test, 2 sided; Independent t-test of change values

12. Secondary Outcome: Body Mass Index
Description: (body mass) divided by (height x height)
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
kg/m^2
  Week 0 | 22.7 (3.7) | 22.8 (2.5)
  Week 16 | 22.7 (3.7) | 22.9 (2.3)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.9135, t-test, 2 sided; Independent t-test of change values

13. Secondary Outcome: Change in Waist Circumference
Description: Measurement of waist circumference using World Health Organization guidelines
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
cm
  Week 0 | 80.5 (9.6) | 22.9 (2.3)
  Week 16 | 80.4 (9.6) | 22.8 (2.5)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.5859, t-test, 2 sided; Independent t-test of change values

14. Secondary Outcome: Change in Appetite
Description: A subjective visual analogue scale consisting of a 100 mm line for each term (1) hunger; (2) fullness; (3) desire to eat; (4) prospective food consumption. Subjects respond by placing a mark on the line that is anchored with an extreme answer at either end (e.g. "not felt at all" and "felt the greatest")
  A composite appetite score is computed by: (hunger + desire to eat + (100 - fullness) + prospective food consumption) divided by 4. With a maximum score of 400 for the greatest possible appetite (represented by hunger = 100; desire to eat = 100; fullness = 0 and prospective food consumption = 100) and a minimum score of 0 (represented by hunger = 0; desire to eat = 0; fullness = 100 and prospective food consumption = 0)
Time Frame: Assessed at week 0, week 4, week 8, week 12 and week 16, week 0 and 16 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
score on a scale
  Week 0 | 215 (17) | 209 (64)
  Week 16 | 194 (104) | 185 (81)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.9379, t-test, 2 sided; Independent t-test of change values

15. Secondary Outcome: Dietary Carotenoids
Description: Analysis of dietary carotenoids using 3-day food records
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
ug
  Week 0 | 8627.1 (1637.1) | 11087.4 (1708.3)
  Week 16 | 10487.8 (1099.5) | 12845.98 (1791.12)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.9717, t-test, 2 sided; t-test of change values

16. Secondary Outcome: Change in Sleep Quality
Description: Measured using The Pittsburgh Sleep Quality Index (PSQI) and sleep evaluation questionnaire
Time Frame: Pre- and post-intervention (Week 16)
Reporting Status: Not Posted, anticipated posting 2020-09

17. Secondary Outcome: Change in Cognitive Function
Description: Measured using Montreal cognitive assessment (MOCA)
Time Frame: Pre- and post-intervention (Week 16)
Reporting Status: Not Posted, anticipated posting 2020-09

18. Primary Outcome: Change in Plasma Endothelin-1
Description: Concentrations of plasma endothelin-1 using commercially available ELISA assay kits.
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
pg/mL
  Endothelin1 Week 0 | 1.31 (0.56) | 1.19 (0.6)
  Endothelin1 Week 16 | 1.11 (0.48) | 1.04 (0.51)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.7052, t-test, 2 sided; Independent t-test of change values
Statistical Analysis 2: Comparison: Healthy Diet; Test type: Superiority; p = 0.07, t-test, 2 sided; Paired t-test between Week 0 and Week 16 endothelin-1 concentrations
Statistical Analysis 3: Comparison: Wolfberry With Healthy Diet; Test type: Superiority; p = 0.005, t-test, 2 sided — Paired t-test between Week 0 and Week 16 endothelin-1 concentrations

19. Primary Outcome: Change in Plasma ICAM-1
Description: Concentrations of plasma intercellular adhesion molecule-1 using commercially available ELISA assay kits.
Time Frame: Pre- and post-intervention (Week 16)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
Number analyzed (Participants) | 22 | 18
ng/mL
  ICAM-1 Week 0 | 7.4 (2.33) | 7.1 (2.52)
  ICAM-1 Week 16 | 7.43 (2.43) | 7.14 (2.25)
Statistical Analysis 1: Comparison: Wolfberry With Healthy Diet vs Healthy Diet; Test type: Superiority; p = 0.9426, t-test, 2 sided — Independent t-test of change values

ADVERSE EVENTS:
Time Frame: 1 year
Description: There is no known risk associated with the consumption of wolfberry or a healthy eating pattern diet according to earlier intervention studies of a similar nature
Arm/Group | Wolfberry With Healthy Diet | Healthy Diet
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

LIMITATIONS AND CAVEATS:
There are no limitations to this trial currently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03535844/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT03535844/ICF_001.pdf